CLINICAL TRIAL: NCT03847935
Title: Trigger Finger Treatment - An Outcomes Study. Comparing 6 Traditional Treatment Techniques
Brief Title: Trigger Finger Treatment
Status: Completed | Type: Observational
Sponsor: University of Massachusetts, Lowell (Other)
Collaborators: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, ELewis, Associate Professor, University of Massachusetts, Lowell
Other Study IDs: H-12583
Record Dates: First submitted 2019-02-08; First posted 2019-02-20 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Trigger Finger; Trigger Digit; Stenosing Tenosynovitis
Keywords: treatment outcome; hand therapy; physical therapy; occupational therapy
MeSH Terms: conditions — Trigger Finger Disorder; Tendon Entrapment | interventions — Surgical Procedures, Operative; Physical Therapy Modalities; Occupational Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Surgery: Patients who underwent surgical release of A1 pulley
  Interventions: Procedure: surgery
- corticosteroid injections only: Patients who underwent local corticosteroid injections only, and no other treatment
  Interventions: Procedure: corticosteroid injections
- hand therapy only occupational/physical: 1 visit: orthosis fabrication, range of motion, nodule and ice massage.
  Interventions: Other: Hand Therapy
- Injection and Hand therapy: This group of participants received a combination of corticosteroid injection in the affected finger and one visit of hand therapy.
  Interventions: Procedure: corticosteroid injections; Other: Hand Therapy
- Modality Hand Therapy: Ongoing hand therapy treatment, which included the above plus modalities such as ultrasound or iontophoresis.
  Interventions: Other: Modality Hand Therapy
- Injection and Modality Hand Therapy: Ccombination of local cortiscosteroid injection to the affected digit and ongoing hand therapy with modalities.
  Interventions: Procedure: corticosteroid injections; Other: Modality Hand Therapy

INTERVENTIONS:
Procedure: surgery — A1 pulley release of finger
  Groups: Surgery
Procedure: corticosteroid injections — corticosteroid injection to A1 pulley
  Groups: Injection and Hand therapy; Injection and Modality Hand Therapy; corticosteroid injections only
Other: Hand Therapy — orthosis fabrication, therapeutic exercise for range of motion to digits, ice massage, nodule massage, patient education,
  Other Names: physical therapy; occupational therapy
  Groups: Injection and Hand therapy; hand therapy only occupational/physical
Other: Modality Hand Therapy — orthosis fabrication, therapeutic exercise for range of motion to digits, ice massage, nodule massage, patient education, plus modalities such as ultrasound, iontophoresis
  Groups: Injection and Modality Hand Therapy; Modality Hand Therapy

SUMMARY:
Trigger finger is a common disorder of the hand which causes pain at the A1 pulley, inflammation, stiffness and/or snapping during movement. This observational study compared all of the possible treatments and combinations of treatments for trigger finger at the A1 pulley, including surgery, cortisone injections and hand therapy.

DETAILED DESCRIPTION:
Trigger finger is a common disorder of the hand which causes pain at the A1 pulley, inflammation, stiffness or snapping during movement. This can be very debilitating. Current treatment includes local steroid injection, oral NSAIDS, resting orthoses, physical or occupational therapy and surgical intervention. The aim of this prospective study with an observational design was to determine the outcome between surgical, hand therapy rehabilitation, and corticosteroid injection interventions for trigger finger. There were 6 treatment groups: surgery, corticosteroid injection, 1 visit of hand therapy for orthosis fabrication and therapeutic exercise, hand therapy in combination with cortisone injection, Modality hand therapy alone (ongoing visits) or with corticosteroid injections.

ELIGIBILITY:
Inclusion Criteria:

* trigger finger in digit 2-5

Exclusion Criteria:

* if prior treatment for trigger finger, or Trigger thumb

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing medical treatment or hand therapy for trigger finger in digits #2-5 at the hand clinic. Patients were dropped from the study if they had changed to a different treatment.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2007-12-10 (Actual); Primary Completion 2012-12-08 (Actual); Study Completion 2012-12-08 (Actual)

PRIMARY OUTCOMES:
Change in Functional use using Quick DASH 6 weeks | Day 1, 6 weeks
  Change from baseline to 6 weeks Quick DASH
Change in Functional use using Quick DASH 3 months | Day 1, 3 months
  Change from baseline to 3 months Quick DASH
Change in Functional use using Quick DASH 6 months | Day 1, 6 months
  Change from baseline to 6 months Quick DASH
Change in Edema 6 weeks | day 1, 6 weeks
  Baseline to 6 weeks Circumferential measurement in centimeters of the proximal phalanx
Change in Edema 3 months | day 1, 3 months
  Baseline to 3 months weeks Circumferential measurement in centimeters of the proximal phalanx
Change in Edema 6 months | day 1, 6 months
  Baseline to 6 months weeks Circumferential measurement in centimeters of the proximal phalanx
Change in Pain on a likert scale 6 weeks | 1 day, 6 weeks
  Baseline to 6 weeks pain on a 0-10 scale
Change in Pain on a likert scale 3 months | 1 day, 3 months
  Baseline to 3 months pain on a 0-10 scale
Change in Pain on a likert scale 6 months | 1 day, 6 months
  Baseline to 6 months pain on a 0-10 scale
Change in Range of motion 6 weeks | 1 day, 6 weeks
  Baseline to 6 weeks flexion and extension range of motion at metacarpophalangeal (MCP), proximal interphalangeal (PIP) and distal interphalangeal (DIP) using a finger goniometer.
Change in Range of motion 3 months | 1 day, 3 months
  Baseline to 3 months flexion and extension range of motion at metacarpophalangeal (MCP), proximal interphalangeal (PIP) and distal interphalangeal (DIP) using a finger goniometer.
Change in Range of motion 6 months | 1 day, 6 months
  Baseline to 6 months flexion and extension range of motion at metacarpophalangeal (MCP), proximal interphalangeal (PIP) and distal interphalangeal (DIP) using a finger goniometer.
Change in Severity or Grade of triggering 6 weeks | 1 day, 6 weeks
  Baseline to 6 weeks Using the scale by Patel and Bassini to measure the amount of triggering 1=normal joint, 6=locked in flexion
Change in Severity or Grade of triggering 3 months | 1 day, 3 months
  Baseline to 3 months Using the scale by Patel and Bassini to measure the amount of triggering 1=normal joint, 6=locked in flexion
Change in Severity or Grade of triggering 6 months | 1 day, 6 months
  Baseline to 6 months Using the scale by Patel and Bassini to measure the amount of triggering 1=normal joint, 6=locked in flexion

CONTACTS AND LOCATIONS:
Overall Officials: Erika S. Lewis, Ed.D, Principal Investigator — Associate Professor, University of Massachusetts Lowell

IPD SHARING:
Plan to Share IPD: No
There are no plans for sharing the IPD

REFERENCES:
- [Background] Lewis E, Fors L, Tharion WJ. Interrater and intrarater reliability of finger goniometric measurements. Am J Occup Ther. 2010 Jul-Aug;64(4):555-61. doi: 10.5014/ajot.2010.09028. PMID 20825126